CLINICAL TRIAL: NCT04734119
Title: Patient Satisfaction With Perioperative Anesthetic Care: Is Continuity of Care Crucial?
Brief Title: Patient Satisfaction With Perioperative Anesthetic Care
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr., Meir Medical Center
Other Study IDs: 0226-18-MMC
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Anesthesia
Keywords: anesthesia; patient satisfaction; continuity of care
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A- same anesthesiologist: In Group A patients were evaluated preoperatively and anesthetized by the same anesthesiologist.
  Interventions: Other: Pre operative evaluation and anesthesia administration by the same anesthesiologist
- Group B- different anesthesiologist: In Group B the preoperative assessment and actual anesthesia was performed by two different anesthesiologists

INTERVENTIONS:
Other: Pre operative evaluation and anesthesia administration by the same anesthesiologist — Pre operative evaluation and anesthesia administration by the same anesthesiologist (instead of two different anesthesiologists, as routinely performed in our medical center)
  Groups: Group A- same anesthesiologist

SUMMARY:
The doctor-patient relationship, medical competence and patient expectations influence patient satisfaction with anesthesia. Preoperatively all patients are routinely assessed by an anesthesiologist. However, in many centers, the anesthesiologist who performs the preoperative evaluation will not necessarily be the anesthesiologist who provides the intraoperative service. This study evaluated the effect of this practice on patient satisfaction, level of confidence and anxiety among adult patients undergoing elective surgery.

DETAILED DESCRIPTION:
Background: The doctor-patient relationship, medical competence and patient expectations influence patient satisfaction with anesthesia. Preoperatively all patients are routinely assessed by an anesthesiologist. However, in many centers, the anesthesiologist who performs the preoperative evaluation will not necessarily be the anesthesiologist who provides the intraoperative service. This study evaluated the effect of this practice on patient satisfaction, level of confidence and anxiety among adult patients undergoing elective surgery.

Methods: 100 patients scheduled for elective surgery under general anesthesia were randomly divided into 2 equal groups: In Group A patients were evaluated and anesthetized by the same anesthesiologist. In Group B the preoperative assessment and actual anesthesia was performed by two different anesthesiologists. On the first postoperative day all patients completed a questionnaire designed to evaluate their sense of preoperative security (confidence) and their overall satisfaction with the anesthetic experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under general anesthesia
* Period- 12.2018-03.2019
* ASA score 1 to3
* Hebrew is the patient mother tongue
* The patient was pre-operatively evaluated by an anesthesiologist at least one day before surgery
* Duration of surgery is more than 1 hour
* The anesthesiologist has more than 2 years experience at work

Exclusion Criteria:

* The patient suffers from severe cognitive decline or severe psychiatric illness
* The patient is unable to answer the questionnaire by himself/herself
* The patient received pre-operative sedation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery under general anesthesia between 12.2018 and 03.2019
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Level of patient satisfaction | Post operative day 1
  Level of patient satisfaction from anesthesia management, as described by patient questionnaire, ranked 1-5 (1- very satisfied, 5- not satisfied at all).

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center Kfar Saba, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No